CLINICAL TRIAL: NCT04264611
Title: Effects of Short Foot and Towel Curl Exercises on Foot Arches Morphology, Dynamic and Static Pedobarographic Parameters and Balance: Randomized Controlled Trial
Brief Title: Comparing the Effects of Foot Core Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Collaborators: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, MERVE SEVİK, Research Assistant, Physical Therapist, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 170054
Record Dates: First submitted 2020-02-07; First posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Foot Injuries and Disorders; Balance; Distorted
Keywords: Foot Core System; Plantar Intrinsic Foot Muscles; Short Foot Exercise; Towel Curl Exercise; Medial Longitudinal Arch; Pedobarography;; Balance
MeSH Terms: conditions — Foot Injuries; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Short Foot Exercise Group (Experimental): The group that received the short foot exercise
  Interventions: Other: Experimental: Short Foot Exercise Group
- Towel Curl Exercise Group (Experimental): The group that received the towel curl exercise
  Interventions: Other: Experimental: Towel Curl Exercise Group
- Control Group (No Intervention): The group that received no exercise

INTERVENTIONS:
Other: Experimental: Short Foot Exercise Group — Short foot exercise which was performed under the supervision of physiotherapist for four weeks in 30 repetitions five days a week.
  Arms: Short Foot Exercise Group
Other: Experimental: Towel Curl Exercise Group — Towel curl exercise which was performed under the supervision of physiotherapist for four weeks in 30 repetitions five days a week.
  Arms: Towel Curl Exercise Group

SUMMARY:
The purpose of the study was to compare the effects of towel curl exercises and short foot exercises on pedobarographic parameters and balance. 91 healthy students (63 females, 28 males) with mean age of 20,65±2,41 years who attend to Muğla Sıtkı Koçman University, Faculty of Health Sciences and met the inclusion criteria and volunteered to participate included in this randomized controlled study. Participants were randomly divided into, Short Foot Exercise(n=28), Towel Curl Exercise (n=31) and Control Groups (n=32). Participant's demographic information were recorded, foot number measurement, navicular drop test, metatarsal width measurement, static and dynamic pedobarographic evaluations, and the balance evaluation were performed. Following the initial assessment, participants who included in Short Foot and Towel Curl Exercise Group performed the exercises that they were assigned to under the supervision of a physiotherapist for 4 weeks and no exercise was given to the control group. After the completion of 4 weeks all the initial assessments were repeated in all groups.

DETAILED DESCRIPTION:
This study was planned as a randomized controlled study to compare the effects of Towel Curl Exercise (TCE) which is often used in physiotherapy clinics for injuries caused by contractile structures of the foot, especially in cases of pes planus and Short Foot Exercise (SFE) which has increasing popularity with recent studies. This study was conducted between March 2018 and June 2018. Firstly, informed consent form was signed by participants and that the rights of the subjects were protected. The participants were randomized using a computer assisted randomization method; they were divided into Short Foot Exercise Group (SFEG), Towel Curl Exercise Group (TCEG) and Control Group (CG). Pre and post-test design was used for this randomized controlled study. The dependent variables recorded before and after four weeks of SFE and TCE were; changes in navicular drop, metatarsal enlargement amounts, static and dynamic pedobarographic parameters and balance scores. Evaluations and exercises of the individuals were performed by the same researcher physiotherapist. The study protocol was approved by the ethics committee of Mugla Sıtkı Koçman University (Protocol no: 170054).

Subjects The study was conducted on 91 healthy subjects, 68 female and 23 male, with a mean age of 20.65 ± 2.410 years (18 to 34 years). Four of SFEG, three of TCEG, four of CG patients had left dominant feet and the others had right dominant feet.

Procedures Subjects were invited for evaluation in clinic for three consecutive days; first day their age, height, weight values, foot sizes, navicular drop distance (ND) and metatarsal width (MTW) were measured and determined their dominant lower extremity. Balance scores were recorded with SportKat device on the second day and static and dynamic pedobarography results recorded on the third day. Navicular drop test was used to evaluate the flexibility of the foot. In this study, MTW were measured in order to evaluate the effects of SFE and TCE on the flexibility of fore foot. Diagnostic Support Electronic Baropodometer and Milletrix software (DIASU®, Italy) were used for static and dynamic pedobarographic measurements to evaluate foot plantar pressure distribution.

After all evaluations had been completed the exercises were taught by the researcher physiotherapist with video and verbal narration and exercise were tested on each participant who were included Short Foot Exercise Group and Towel Curl Exercise Group.

Subjects who completed all evaluations, started their exercises according to the exercise groups they were assigned to and the CG was not given any exercise. Exercises were performed under the supervision of physiotherapist for four weeks in 30 repetitions five days a week. Exercises were progressed by sitting for one week, standing on double leg in the 2nd week and standing on one leg in the 3rd and 4th weeks in both groups. The individuals in the control group were asked not to go out of their daily physical activity routine during this four-week period.

The SFEG, TCEG and CG were called to the clinic again and their final measurements were recorded after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Be over 18 years old
* Sign informed consent form
* Have not experienced towel curl exercise and short foot exercise

Exclusion Criteria:

* Any sign of foot pain
* The presence of problems affecting the foot such as diagnosed patellofemoral pain syndrome, plantar fasciitis, anterior or posterior tibialis dysfunction
* In the last 6 months; presence of injury or surgical operation of the lower extremity
* Lower limb length inequalities that affect gait
* The presence of a systemic, neurological, orthopedic disease or deformity that will affect motor function, balance and gait

Ages: 18 Years to 34 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Measuring navicular drop distance | 3 minutes
  The individual was placed on a stool with the bare foot, hip, knee and ankle flexed 90 degrees with the foot in full contact with the floor and was asked to look at a fixed point opposite. In this position the navicular tubercle was determined with the erasable pen and the navicular height above the ground was marked on an index card. Then, the individual was asked to stand up without changing the position of her/his heels and while standing, the navicular tubercle was again determined and its height above the ground was marked on the index card. The distance between the navicular heights marked on the index card in the sitting and standing positions was measured with the help of the INSIZE® 1108-200 digital caliper and recorded as navicular drop distance in mm.
Measuring metatarsal width | 3 minutes
  Metatarsal width was recorded by measuring the extreme distance between the medial soft tissue line at the first metatarsal head level and the lateral soft tissue line at the fifth metatarsal head level. It was measured using the INSIZE® 1108-200 digital caliper for both feet while giving equal weight to both lower extremities in the sitting position at 90 degrees flexion of the hip, knee and ankle joints and giving equal weight to both lower extremities in the standing position. Metatarsal width in sitting and standing positions were recorded and the difference between them was calculated and recorded as the amount of metatarsal enlargement in mm.
Pedobarographic evaluation | 10 minutes
  Diagnostic Support Electronic Baropodometer and Milletrix software (DIASU®, Italy) were used for static and dynamic pedobarographic measurements to evaluate foot plantar pressure distrubution. Static measurements were made with the patient standing on a platform with pressure sensor, with two bare feet, in a loose standing position, looking at a fixed point opposite. The dynamic measurements were made after the individuals performed a trial walk on the platform once. Individuals were asked to walk self- selected speed and pattern. The average values of 4 dynamic measurements were taken for both foot and the results were recorded.
Balance evaluation | 10 minutes
  Static and dynamic balances of individuals on double and single legs were evaluated using SportKAT® Model 650-TS, LLC, USA. The monitor was positioned 130 cm forward and at the eye level of the subject. Individuals standing on the platform whose pressure was set to 6 PSI and they were asked to position their arms across the shoulders. The test was canceled and repeated in the event that individuals arms were distorted or they fall off the platform.

SECONDARY OUTCOMES:
Foot size | 1 minute
  Foot size was measured using ruler which is proper for Turkey and European standarts.

CONTACTS AND LOCATIONS:
Locations (1):
- Lokman Hekim University, Ankara, Çankaya, Turkey (Türkiye)